CLINICAL TRIAL: NCT00631371
Title: Phase 3b, Randomized, Open-Label Study Of Bevacizumab + Temsirolimus Vs. Bevacizumab + Interferon-Alfa As First-Line Treatment In Subjects With Advanced Renal Cell Carcinoma
Brief Title: Study Comparing Bevacizumab + Temsirolimus vs. Bevacizumab + Interferon-Alfa In Advanced Renal Cell Carcinoma Subjects
Acronym: INTORACT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3066K1-3311; B1771006 (Other: Alias Study Number); 2007-003793-26 (EudraCT Number)
Record Dates: First submitted 2008-02-28; First posted 2008-03-07 (Estimated); Results first posted 2013-06-04 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-03

CONDITIONS: Renal Cell Carcinoma
Keywords: temsirolimus; renal cell carcinoma; kidney cancer; urogenital cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms; Urogenital Neoplasms | interventions — Bevacizumab; temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Bevacizumab 10 mg/kg intravenous (IV) q8wks + Temsirolimus 25 mg IV weekly
  Interventions: Drug: Bevacizumab; Drug: Temsirolimus
- 2 (Active Comparator): Bevacizumab 10 mg/kg intravenous (IV) q8wks + Interferon-Alfa 9MU SC TIW
  Interventions: Drug: Bevacizumab; Drug: Interferon-Alfa 9MU

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab 10 mg/kg intravenous (IV) q8wks
  Other Names: Torisel
  Arms: 1
Drug: Temsirolimus — Temsirolimus 25 mg IV weekly
  Arms: 1
Drug: Bevacizumab — Bevacizumab 10 mg/kg intravenous (IV) q8wks
  Arms: 2
Drug: Interferon-Alfa 9MU — Interferon-Alfa 9MU SC TIW
  Arms: 2

SUMMARY:
Primary objective: Comparison of independently assessed progression free survival (PFS) in subjects administered Bevacizumab + Temsirolimus vs. those administered Bevacizumab + Interferon-Alfa. Secondary objectives: safety, Investigator assessed PFS, objective response rate (independently assessed), and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Histologically and/or cytologically confirmed to have advanced renal cell carcinoma (RCC)
* Majority component of conventional clear-cell type is mandatory
* At least 1 measurable lesion (per RECIST)

Exclusion Criteria:

* Prior systemic treatment for RCC
* Evidence of current or prior central nervous system (CNS) metastases
* Cardiovascular disease
* Pregnant or nursing women
* Additional criteria applies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 791 (Actual)
Dates: Start 2008-04; Primary Completion 2012-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (171):
- United States (24):
  - Hematology Oncology Services of Arkansas, Little Rock, Arkansas
  - South County Hematology/Oncology, Chula Vista, California
  - Cancer Center Oncology Medical Group, La Mesa, California
  - UCLA Medical Center, Los Angeles, California
  - UCLA, Los Angeles, California
  - North County Oncology Medical Clinic, Oceanside, California
  - Medical Oncology Associates - SD, San Diego, California
  - Sharp Memorial Hospital Investigational Pharmacy, San Diego, California
  - Sharp Rees-Stealy, San Diego, California
  - California Pacific Medical Center, San Francisco, California
  - Pacific Hematology/Oncology Associates, San Francisco, California
  - San Francisco Oncology Associates, San Francisco, California
  - Cohen & Hufford MD's INC, San Francisco, California
  - The Jones Clinic, PC, New Albany, Mississippi
  - The Cleveland Clinic, Cleveland, Ohio
  - Edmond Oncology Center, Edmond, Oklahoma
  - OU Medical Center, Oklahoma City, Oklahoma
  - OU Physician's Building, Oklahoma City, Oklahoma
  - University of Oklahoma, Oklahoma City, Oklahoma
  - The Jones Clinic, PC, Germantown, Tennessee
  - The Vanderbilt Clinic, Nashville, Tennessee
  - University of Washington Medical Center, Seattle, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
- Argentina (3):
  - Centro Oncológico Rosario, Rosario, Santa Fe Province
  - ISIS Clinica Especializado, Santa Fe, Santa Fe Province
  - Centro Medico San Roque, San Miguel de Tucumán, Tucumán Province
- Australia (5):
  - Mater Adult Hospital, South Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Ashford Cancer Center Research, Kurralta Park, South Australia
  - Cancer Care SA, Kurralta Park
  - Mater Private Hospital, South Brisbane
- Belgium (4):
  - ZNA Middelheim, Antwerp
  - Universitair Ziekenhuis Gent, Ghent
  - Jessa Ziekenhuis - campus Virga Jessa, Hasselt
  - Cliniques Universitaires de Mont-Godinne UCL, Mont-Godinne
- Brazil (13):
  - Centro Goiano de Oncologia, Goiânia, Goiás
  - Centro Goiano de Oncologia - CGO, Goiânia, Goiás
  - ProCura - Centro Goiano de Pesquisa Clínica Ltda, Goiânia, Goiás
  - Instituto Nacional de Cancer - INCA, Rio de Janeiro, Rio de Janeiro
  - Instituto Nacional do Cancer - INCA, Rio de Janeiro, Rio de Janeiro
  - Associaçao Hospital de Caridade Ijui, Ijuí, Rio Grande do Sul
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Clinica de Oncologia de Porto Alegre - Sociedade Simples Ltda., Porto Alegre, Rio Grande do Sul
  - Clínica de Oncologia de Porto Alegre Sociedade Simples Ltda, Porto Alegre, Rio Grande do Sul
  - Fundação Pio XII - Hospital de Câncer de Barretos, Barretos, São Paulo
  - Instituto de Oncologia de Piracicaba S/S Ltda, Piracicaba, São Paulo
  - Instituto do Cancer do Estado de Sao Paulo Octavio Frias de Oliveira - ICESP, São Paulo, São Paulo
  - Irmandade da Santa Casa de Misericordia de Porto Alegre, Porto Alegre
- Canada (2):
  - Odette Cancer Centre, Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Centre de Sante et de Services Sociaux de Rimouski - Neigette, Rimouski, Quebec
- Chile (3):
  - Instituto Clinico Oncologico del Sur, Santiago, Chile
  - Instituto Nacional del Cancer, Santiago, Region Metropolitana / Chile
  - Fundacion Arturo Lopez Perez, Santiago
- Oncologos del Occidente S.A, Pereira, Risaralda Department, Colombia
- Czechia (4):
  - Oblastni nemocnice Jicin a s, Jičín, Ceska Republika
  - Masarykuv onkologicky ustav, Brno
  - Fakultni nemocnice Olomouc, Olomouc
  - Krajska zdravotni, a.s., Ústí nad Labem
- France (9):
  - Centre Jean Perrin, Clermont-Ferrand
  - Clinique Sainte Marguerite, Hyères
  - Hopital Andre Mignot, Le Chesnay
  - Centre médical Oncogard, Nîmes
  - CHU de Poitiers, Poitiers
  - CHU de Rouen, Rouen
  - Centre rené Gauducheau, Saint-Herblain-Nantes
  - Hopital Foch, Suresnes
  - Institut Gustave Roussy, Villejuif
- Germany (4):
  - Vivantes Klinikum am Urban, Neztwerk fuer Gesundheit GmbH, Berlin
  - Universitaetsklinikum Hamburg Eppendorf, Hamburg
  - Klinikum Region Hannover, Krankenhaus Siloah, Hanover
  - TU Muenchen, rechts der Isar, München
- Hong Kong (3):
  - Prince of Wales Hospital, Hong Kong, Hong Kong
  - Pamela Youde Nethersole Eastern Hospital, Chai Wan
  - Queen Mary Hospital, Hong Kong
- Hungary (6):
  - Orszagos Onkologiai Intezet, Budapest
  - Uzsoki Utcai Korhaz, Budapest
  - Petz Aladar Megyei Oktato Korhaz, Győr
  - Josa Andras Oktato Korhaz Nonprofit Kft., Nyíregyháza
  - Szegedi Tudomanyegyetem, Urologiai Klinika, Szeged
  - Veszprem Megyei Csolnoky Ferenc, Veszprém
- India (10):
  - Vedanta Institute of Medical Sciences, Ahmedabad, Gujarat
  - Healthcare Global Enterprises Limited, Bangalore, Karnataka
  - Lakeshore Hospital & Research Center Limited, Kochi, Kerala
  - Jawaharlal Nehru Cancer Hospital, Department of Medical Oncology, Bhopal, Madhya Pradesh
  - Tata Memorial Center, Mumbai, Maharashtra
  - Tata Memorial Centre, Navi Mumbai, Maharashtra
  - Jehangir Hospital, Pune, Maharashtra
  - Searoc Cancer Centre, Jaipur, Rajasthan
  - Apollo Hospital, Chennai, Tamil Nadu
  - Regional Cancer Centre, Kerela, Trivandrum
- Italy (7):
  - Divisione di Urologia, Azienda Ospedaliera Policlinico Consorziale di Bari, Bari
  - Sezione di Oncologia Medica Centro di Ricerca Clinica, Chieti
  - Unità Operativa di Oncologia, Azienda Ospedaliera Policlinico di Modena, Modena
  - Farmacia del Comitato Etico Provinciale di Modena, Modena
  - Struttura Complessa di Oncologia Medica Ospedale Santa Maria della Misericordia, Perugia
  - IFO- Istituti Fisioterapici Ospitalieri, Roma
  - Azienda Ospedaliera S. Maria, Terni
- University Malaya Medical Centre, Kuala Lumpur, Malaysia, Malaysia
- Hospital Aranda de la Parra, León, Guanajuato, Mexico
- Spaarne Ziekenhuis, Hoofddorp, Netherlands
- Poland (9):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Szpital Specjalistyczny im. L. Rydygiera Sp. z o.o., Krakow
  - Centrum Onkologii Ziemi Lubelskiej im. sw Jana z Dukli, Lublin
  - Szpital Kliniczny Przemienienia Panskiego UM im. Karola Marcinkowskiego w Poznaniu, Poznan
  - Centrum Onkologii, Instytut im. M. Sklodowskiej-Curie, Warsaw
  - Centrum Medyczne Ostrobramska NZOZ "Magodent", Warsaw
  - Wojskowy Instytut Medyczny, Pracownia Badan Cynnosciowych Ukladu Oddechowego, Klinika Chorob Wewnetr, Warsaw
  - Wojskowy Intsytut Medyczny, Zaklad Diagnostyki Laboratoryjnej CSK MON, Warsaw
  - Wojskowy Intsytut Medyczny, Zaklad Medycyny Nuklearnej CSK MON, Warsaw
- Portugal (2):
  - Hospital de San Joao, Porto
  - Hospital de São João, Porto
- Russia (11):
  - Medical Radiology Research Center of the Minzdravsotsrazvitiya of Russia, Obninsk, Kaluga Oblast
  - Leningrad Regional Oncology Dispensary, Saint-Petersburg, Leningradskaya Oblast'
  - Republican Clinical Oncology Dispensary of Minzdrav of Tatarstan Republic, Kazan'
  - Chair of Radiology and Radiotherapy, Moscow
  - N.N. Blokhin Russian Cancer Research Center, Department of Clinical Pharmacology and Chemotherapy, Moscow
  - N.N. Blokhin Russian Cancer Research Center, Department of Urology, Moscow
  - Moscow Scientific Research Oncology Institute P.A. Herzen, Moscow
  - Privolzhskiy District Medical Center of Federal Biomedical Agency, Nizhny Novgorod
  - Scientific research Institute of Oncology N.N. Petrov, Pesochny, Saint-Petersburg
  - City Hospital No.26, Saint Petersburg
  - City Pokrovskaya Hospital, Saint Petersburg
- Serbia (3):
  - Clinical Center of Serbia, Belgrade
  - Institute for Oncology and Radiology of Serbia, Belgrade
  - Military Medical Academy, Belgrade
- National Cancer Centre Singapore, Singapore, Singapore
- Slovakia (11):
  - Fakultna Nemocnica s poliklinikou F D Roosevelta, Banská Bystrica
  - Oddelenie funkcnej diagnostiky, Banská Bystrica
  - Klinika pneumologie a ftiziologie FNsP LFUK, Bratislava
  - Fakultna Nemocnica s poliklinikou akad L Derera, Bratislava
  - Klinica nuklcarncj mediciny, Martin
  - Klinika nuklearnej mediciny JLF UK a Martinskej fakultnej nemocnice, Martin
  - Klinika tuberkulozy a plucnych chorob UK JLF a Martinskej fakultnej nemocince, Martin
  - Nemocnica s poliklinikou Skalica, Skalica
  - KK MED, s.r.o., Žilina
  - MEDIVASA s.r.o., Žilina
  - Nemocnica s poliklinikou Zilina, Žilina
- South Africa (7):
  - GVI Oncology Trial Unit, Kraaifontein, Cape Town
  - Westridge Medical Centre, Mayville, Durban
  - Pretoria Urology Hospital, Hatfield, Pretoria
  - Panorama Medical Centre, Panorama, Cape Town, Western Cape
  - University of the Witwatersrand Oncology, Parktown
  - Langenhoven Drive Oncology Centre, Port Elizabeth
  - Dr. Fourie & Voges, Pretoria
- South Korea (2):
  - Samsung Medical Center, Seoul, Korea
  - Yonsei University Health System-Severance Hospital, Seoul
- Spain (6):
  - Hospital Sant Creu I Sant Pau, Barcelona, Barcelona
  - Institut Catala Doncologia, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital de Madrid Norte-Sanchinarro, Madrid, Madrid
  - Hospital del mar de Barcelona, Barcelona
  - Instituto Valenciano de Oncología, Valencia
- Taiwan (5):
  - Veterans General Hospital-Taipei, Taipei, ROC
  - National Taiwan University Hospital, Taipei TOC, Taiwan
  - Tri-Service General Hospital, Neihu District, Tapei
  - China Medical University Hospital, Taichung
  - Division of Oncology, Taoyuan District
- Ukraine (9):
  - Universitet, kafedra onkologyy, Chenivtsi
  - A.P Romodanov Itstitut nejrohirurhii, Chernivtsi
  - Uchbobo-naukovyi likuvalnyi kompleks DDMU im. M.Gor'kogo, Donetsk
  - Donetskyy Oblasyy protypukhlynnyy Tsenter, Donetsk
  - Donetske Obl. clinico-teritorial'ne medichne ob'yednannya, Donetsk
  - "State Institution ""Institute for Occupational Health of the, Kiev
  - R.E.Kavetsky Institute of experimental pathology, oncology and radiobiology NAS of Ukraine,Laborator, Kiev
  - A.P Romodanov Itstitut nejrohirurhii, Kiyv
  - Oblasnyy onkologychnyy dispanser, onkourologichne viddilennya, Ivano-Frankivskiy Derzhavniy Medichni, Medychna Vul., Ivano-Frankivsk
- United Kingdom (4):
  - Southampton General Hospital, Southampton, Hampshire
  - Christie Hospital, Withington, Manchester
  - University of Leeds, Leeds, North Yorkshire
  - Guy's Hospital, London

REFERENCES:
- [Derived] Aldin A, Besiroglu B, Adams A, Monsef I, Piechotta V, Tomlinson E, Hornbach C, Dressen N, Goldkuhle M, Maisch P, Dahm P, Heidenreich A, Skoetz N. First-line therapy for adults with advanced renal cell carcinoma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 May 4;5(5):CD013798. doi: 10.1002/14651858.CD013798.pub2. PMID 37146227
- [Derived] de Velasco G, McKay RR, Lin X, Moreira RB, Simantov R, Choueiri TK. Comprehensive Analysis of Survival Outcomes in Non-Clear Cell Renal Cell Carcinoma Patients Treated in Clinical Trials. Clin Genitourin Cancer. 2017 Dec;15(6):652-660.e1. doi: 10.1016/j.clgc.2017.03.004. Epub 2017 Mar 21. PMID 28410911
- [Derived] Grunwald V, Lin X, Kalanovic D, Simantov R. Early Tumour Shrinkage: A Tool for the Detection of Early Clinical Activity in Metastatic Renal Cell Carcinoma. Eur Urol. 2016 Dec;70(6):1006-1015. doi: 10.1016/j.eururo.2016.05.010. Epub 2016 May 26. PMID 27238653
- [Derived] Rini BI, Bellmunt J, Clancy J, Wang K, Niethammer AG, Hariharan S, Escudier B. Randomized phase III trial of temsirolimus and bevacizumab versus interferon alfa and bevacizumab in metastatic renal cell carcinoma: INTORACT trial. J Clin Oncol. 2014 Mar 10;32(8):752-9. doi: 10.1200/JCO.2013.50.5305. Epub 2013 Dec 2. PMID 24297945
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3066K1-3311&StudyName=Study%20Comparing%20Bevacizumab%20+%20Temsirolimus%20vs.%20Bevacizumab%20+%20Interferon-Alfa%20In%20Advanced%20Renal%20Cell%20Carcinoma%20Subjects

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Approximately 800 participants enrolled in this study at 200 sites.
Pre-assignment Details: Participants were randomized in a 1:1 ratio, stratified by prior nephrectomy status (yes/no) and Memorial Sloan Kettering Cancer Center (MSKCC) risk factors (good/intermediate/poor), and received either the combination treatment of Temisirolimus + Bevacizumab (Temsr+Bev) or Interferon-alfa + Bevacizumab (IFN+Bev).
Groups:
- Bevacizumab+Temsirolimus: Bevacizumab 10 milligram per kilogram (mg/kg) intravenous infusion over 90 minutes, 60 minutes or 30 minutes depending on the participant's tolerability every other week along with temsirolimus 25 mg intravenous infusion over at least 30 minutes once a week. Treatment was continued until disease progression, unacceptable toxicities, withdrawal of consent, or death.
- Bevacizumab+ Interferon-Alfa: Bevacizumab 10 mg/kg intravenous infusion over 90 minutes, 60 minutes or 30 minutes depending on the participant's tolerability every other week along with interferon-alfa (IFN) 9 million units (MU) subcutaneous injection every 3 times a week. Treatment was continued until disease progression, unacceptable toxicities, withdrawal of consent, or death.
Period: Overall Study
Arm/Group | Bevacizumab+Temsirolimus | Bevacizumab+ Interferon-Alfa
Started | 400 | 391
Treated | 393 | 391
Completed | 0 | 0
Not Completed | 400 | 391
Not completed — Lost to Follow-up | 24 | 19
Not completed — Other reason | 5 | 12
Not completed — subject request | 38 | 45
Not completed — Discontinuation of study by Sponsor | 70 | 76
Not completed — Death | 263 | 239

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bevacizumab+Temsirolimus | Bevacizumab+ Interferon-Alfa | Total
Number analyzed (Participants) | 400 | 391 | 791
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (10.1) | 58.2 (10.4) | 58.4 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114 | 121 | 235
  Male | 286 | 270 | 556

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS): Independent-Assessment
Description: PFS was defined as the interval from the date of randomization until the earlier date of progression or death. Progression was assessed by independent imaging reviewers using Response Evaluation Criteria in Solid Tumors (RECIST) criteria which is 20% increase in sum of longest diameter of target lesions from nadir (the lowest blood counts); measurable increase in non-target lesion; appearance of new lesions.
Time Frame: Baseline until disease progression, initiation of new anticancer treatment, or death, assessed every 8 weeks (up to cut-off date: 19 April 2012)
Population: Intent-to-treat (ITT) population included all participants who were randomized to the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab+Temsirolimus | Bevacizumab+ Interferon-Alfa
Number analyzed (Participants) | 400 | 391
months | 9.1 [8.1 to 10.2] | 9.3 [9.0 to 11.2]
Statistical Analysis 1: Comparison: Bevacizumab+Temsirolimus vs Bevacizumab+ Interferon-Alfa; P value was based on 1-sided stratified log-rank test (stratification factors: prior nephrectomy [yes/no] and Memorial Sloan Kettering Cancer Center [MSKCC] risk factors [good/intermediate/poor] at time of randomization). The hazard ratio and corresponding 95 percent (%) confidence interval (CI) from the stratified cox proportional hazard model were also presented; Test type: Superiority or Other; p = 0.8, Log Rank; Hazard Ratio (HR) = 1.1, 95% CI 2-sided [0.9 to 1.3]

2. Secondary Outcome: Progression-Free Survival (PFS): Investigator-Assessment
Description: PFS was defined as the interval from the date of randomization until the earlier date of progression or death. Progression was assessed by investigator imaging reviewers using RECIST criteria which is 20% increase in sum of longest diameter of target lesions from nadir (the lowest blood counts); measurable increase in non-target lesion; appearance of new lesions.
Time Frame: as for outcome 1
Population: ITT population included all participants who were randomized to the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab+Temsirolimus | Bevacizumab+ Interferon-Alfa
Number analyzed (Participants) | 400 | 391
months | 9.1 [8.1 to 10.5] | 10.8 [9.1 to 11.2]
Statistical Analysis 1: Comparison: Bevacizumab+Temsirolimus vs Bevacizumab+ Interferon-Alfa; P-value was based on 1-sided stratified log-rank test (stratification factors: prior nephrectomy [yes/no] and MSKCC risk factors [good/intermediate/poor] at time of randomization). The hazard ratio and corresponding 95% CI from the stratified cox proportional hazard model were also presented; Test type: Superiority or Other; p = 0.9, Log Rank; Hazard Ratio (HR) = 1.1, 95% CI 2-sided [1.0 to 1.4]

3. Secondary Outcome: Percentage of Participants With Objective Response (Complete Response/Partial Response): Independent-Assessment
Description: Percentage of participants with OR based assessment of confirmed complete response (CR) or confirmed partial response (PR) according to RECIST. Confirmed response were those that persisted on repeat imaging study at least 4 weeks after initial documentation of response. CR was defined as disappearance of all lesions (target and/or non target). PR were those with at least 30% decrease in sum of the longest dimensions of target lesions taking as a reference the baseline sum longest dimensions, with non target lesions not increased or absent.
Time Frame: as for outcome 1
Population: ITT population included all participants who were randomized to the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab+Temsirolimus | Bevacizumab+ Interferon-Alfa
Number analyzed (Participants) | 400 | 391
percentage of participants | 27.0 [22.7 to 31.6] | 27.4 [23.0 to 32.1]
Statistical Analysis 1: Comparison: Bevacizumab+Temsirolimus vs Bevacizumab+ Interferon-Alfa; P-value (2-sided), risk ratio and associated 95% CI were based on Cochran-Mantel-Haenszel test stratified by prior nephrectomy and MSKCC risk group as randomized; Test type: Superiority or Other; p = 1.0, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.0, 95% CI 2-sided [0.8 to 1.3]

4. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death due to any cause, censored at the last date known alive. Death was determined from adverse event data (where outcome was death) or from follow-up contact data (where the participant current status was death).
Time Frame: Baseline until death due to any cause, assessed every 8 weeks (up to cut-off date: 19 April 2012)
Population: ITT population included all participants who were randomized to the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab+Temsirolimus | Bevacizumab+ Interferon-Alfa
Number analyzed (Participants) | 400 | 391
months | 25.8 [21.1 to 30.7] | 25.5 [22.4 to 30.8]
Statistical Analysis 1: Comparison: Bevacizumab+Temsirolimus vs Bevacizumab+ Interferon-Alfa; P value was based on 1-sided stratified log-rank test (stratification factors: prior nephrectomy [yes/no] and MSKCC risk factors [good/intermediate/poor] at time of randomization). The hazard ratio and corresponding 95% CI from the stratified cox proportional hazard model were also presented; Test type: Superiority or Other; p = 0.6, Log Rank; Hazard Ratio (HR) = 1.0, 95% CI 2-sided [0.9 to 1.3]

ADVERSE EVENTS:
Time Frame: Adverse events were collected and reported from the signing of the informed consent until end of treatment but no later than 30 days after the last dose of study medication.
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Bevacizumab+Temsirolimus | Bevacizumab+ Interferon-Alfa
Serious Adverse Events (participants affected / at risk) | 184/393 | 158/391
Other Adverse Events (participants affected / at risk) | 383/393 | 378/391
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab+Temsirolimus (N=393) | Bevacizumab+ Interferon-Alfa (N=391)
Anaemia (Blood and lymphatic system disorders) | 10 | 12
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 3 | 0
Cardiac valve disease (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0
Coronary ostial stenosis (Cardiac disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Retinopathy (Eye disorders) | 0 | 2
Vitreous floaters (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 8 | 6
Anal fissure (Gastrointestinal disorders) | 2 | 0
Anal fistula (Gastrointestinal disorders) | 2 | 2
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 7 | 5
Gastric fistula (Gastrointestinal disorders) | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 2 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Ileal perforation (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 1
Ileus paralytic (Gastrointestinal disorders) | 1 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 1
Large intestine perforation (Gastrointestinal disorders) | 2 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Painful defaecation (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 2
Pancreatitis acute (Gastrointestinal disorders) | 1 | 1
Proctitis (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 1
Subileus (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 7 | 2
Asthenia (General disorders) | 4 | 5
Chills (General disorders) | 0 | 1
Death (General disorders) | 0 | 4
Disease progression (General disorders) | 13 | 16
Fatigue (General disorders) | 1 | 7
General physical health deterioration (General disorders) | 2 | 6
Injury associated with device (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 5 | 0
Multi-organ failure (General disorders) | 2 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Pain (General disorders) | 1 | 2
Pyrexia (General disorders) | 9 | 7
Sudden death (General disorders) | 5 | 0
Acute hepatic failure (Hepatobiliary disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 3 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Hepatitis toxic (Hepatobiliary disorders) | 0 | 1
Contrast media allergy (Immune system disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0
Abdominal abscess (Infections and infestations) | 0 | 1
Abscess (Infections and infestations) | 0 | 1
Abscess intestinal (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 5 | 2
Anorectal cellulitis (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 0 | 1
Bronchopneumonia (Infections and infestations) | 3 | 1
Cellulitis (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 0 | 1
Diarrhoea infectious (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0
Gangrene (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1
Haematoma infection (Infections and infestations) | 0 | 1
Haemorrhoid infection (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 1
Infectious pleural effusion (Infections and infestations) | 2 | 0
Injection site infection (Infections and infestations) | 0 | 1
Liver abscess (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 1
Lung abscess (Infections and infestations) | 2 | 0
Osteomyelitis chronic (Infections and infestations) | 1 | 0
Perirectal abscess (Infections and infestations) | 2 | 0
Peritoneal abscess (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 3 | 2
Pharyngitis (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 16 | 5
Post procedural infection (Infections and infestations) | 0 | 1
Rectal abscess (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 2 | 1
Scrotal abscess (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 2 | 4
Septic shock (Infections and infestations) | 1 | 2
Sinusitis (Infections and infestations) | 2 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 1
Tooth infection (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 5 | 4
Urosepsis (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Viral pharyngitis (Infections and infestations) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0
Post procedural fistula (Injury, poisoning and procedural complications) | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 2
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 0 | 1
Blood pressure systolic decreased (Investigations) | 1 | 0
Fibrin D dimer increased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 2
Protein urine present (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 3 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 2
Hypophagia (Metabolism and nutrition disorders) | 1 | 0
Ketosis (Metabolism and nutrition disorders) | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Bone lesion (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain stem infarction (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 2
Cerebrovascular accident (Nervous system disorders) | 0 | 3
Dizziness (Nervous system disorders) | 1 | 1
Epilepsy (Nervous system disorders) | 1 | 1
Facial paresis (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 4 | 2
Hypertensive encephalopathy (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1
Mental impairment (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 0 | 4
Transient ischaemic attack (Nervous system disorders) | 0 | 4
Tremor (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 2 | 3
Nephrectasia (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Nephrotic syndrome (Renal and urinary disorders) | 4 | 2
Proteinuria (Renal and urinary disorders) | 2 | 3
Renal disorder (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 5 | 2
Renal impairment (Renal and urinary disorders) | 1 | 0
Ureteral disorder (Renal and urinary disorders) | 0 | 1
Ureteric obstruction (Renal and urinary disorders) | 1 | 0
Ureteric stenosis (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 10
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal septum disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 1
Malignant tumour excision (Surgical and medical procedures) | 1 | 0
Arteriosclerosis (Vascular disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 1 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 1
Haematoma (Vascular disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 6 | 4
Hypertensive crisis (Vascular disorders) | 1 | 1
Lymphoedema (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 1 | 0
Cardio-Respiratory Arrest (Cardiac disorders) | 0 | 1
Condition Aggravated (General disorders) | 1 | 0
Colonic abscess (Infections and infestations) | 0 | 1
Epididymitis (Infections and infestations) | 0 | 1
Plasmodium Malariae Infection (Infections and infestations) | 1 | 0
Pulmonary Tuberculosis (Infections and infestations) | 1 | 0
Pyelonephritis Acute (Infections and infestations) | 0 | 1
Blood Bilirubin Increased (Investigations) | 1 | 0
Blood Creatinine Increased (Investigations) | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Balance Disorder (Nervous system disorders) | 1 | 0
Central Nervous System Haemorrhage (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 3 | 1
Toxic Encephalopathy (Nervous system disorders) | 0 | 1
Vascular Encephalopathy (Nervous system disorders) | 0 | 1
Completed Suicide (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 4 | 3
Cancer Surgery (Surgical and medical procedures) | 1 | 0
Peripheral Venous Disease (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab+Temsirolimus (N=393) | Bevacizumab+ Interferon-Alfa (N=391)
Anaemia (Blood and lymphatic system disorders) | 80 | 66
Leukopenia (Blood and lymphatic system disorders) | 17 | 40
Lymphopenia (Blood and lymphatic system disorders) | 24 | 38
Neutropenia (Blood and lymphatic system disorders) | 18 | 66
Thrombocytopenia (Blood and lymphatic system disorders) | 50 | 40
Abdominal pain (Gastrointestinal disorders) | 48 | 42
Abdominal pain upper (Gastrointestinal disorders) | 31 | 21
Constipation (Gastrointestinal disorders) | 43 | 48
Diarrhoea (Gastrointestinal disorders) | 126 | 86
Gingival bleeding (Gastrointestinal disorders) | 5 | 21
Haemorrhoids (Gastrointestinal disorders) | 28 | 13
Nausea (Gastrointestinal disorders) | 69 | 78
Stomatitis (Gastrointestinal disorders) | 102 | 39
Toothache (Gastrointestinal disorders) | 37 | 14
Vomiting (Gastrointestinal disorders) | 53 | 53
Asthenia (General disorders) | 95 | 113
Chills (General disorders) | 15 | 44
Fatigue (General disorders) | 92 | 122
Influenza like illness (General disorders) | 14 | 48
Mucosal inflammation (General disorders) | 105 | 40
Oedema peripheral (General disorders) | 67 | 32
Pyrexia (General disorders) | 79 | 154
Upper respiratory tract infection (Infections and infestations) | 20 | 15
Urinary tract infection (Infections and infestations) | 23 | 21
Alanine aminotransferase increased (Investigations) | 38 | 35
Aspartate aminotransferase increased (Investigations) | 33 | 41
Blood creatinine increased (Investigations) | 40 | 25
Weight decreased (Investigations) | 90 | 93
Decreased appetite (Metabolism and nutrition disorders) | 103 | 127
Hypercholesterolaemia (Metabolism and nutrition disorders) | 126 | 39
Hyperglycaemia (Metabolism and nutrition disorders) | 86 | 19
Hyperkalaemia (Metabolism and nutrition disorders) | 29 | 37
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 114 | 82
Hypocalcaemia (Metabolism and nutrition disorders) | 24 | 13
Hypomagnesaemia (Metabolism and nutrition disorders) | 20 | 16
Hyponatraemia (Metabolism and nutrition disorders) | 23 | 21
Hypophosphataemia (Metabolism and nutrition disorders) | 40 | 18
Arthralgia (Musculoskeletal and connective tissue disorders) | 52 | 49
Back pain (Musculoskeletal and connective tissue disorders) | 47 | 53
Bone pain (Musculoskeletal and connective tissue disorders) | 18 | 22
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 27 | 19
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 14 | 28
Myalgia (Musculoskeletal and connective tissue disorders) | 19 | 60
Pain in extremity (Musculoskeletal and connective tissue disorders) | 43 | 35
Dizziness (Nervous system disorders) | 29 | 37
Dysgeusia (Nervous system disorders) | 33 | 21
Headache (Nervous system disorders) | 77 | 82
Anxiety (Psychiatric disorders) | 7 | 21
Depression (Psychiatric disorders) | 11 | 22
Insomnia (Psychiatric disorders) | 28 | 31
Proteinuria (Renal and urinary disorders) | 143 | 111
Cough (Respiratory, thoracic and mediastinal disorders) | 79 | 70
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 13 | 30
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 36 | 49
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 110 | 82
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 28 | 16
Dry skin (Skin and subcutaneous tissue disorders) | 27 | 13
Pruritus (Skin and subcutaneous tissue disorders) | 60 | 26
Rash (Skin and subcutaneous tissue disorders) | 126 | 32
Hypertension (Vascular disorders) | 128 | 102
Vertigo (Ear and labyrinth disorders) | 4 | 20
Blood Alkaline Phosphatase Increased (Investigations) | 20 | 14
Hypokalaemia (Metabolism and nutrition disorders) | 20 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.